CLINICAL TRIAL: NCT03889106
Title: Cardiovascular Function and Ribavirin Pharmacokinetics and Pharmacodynamics in Patients With Lassa Fever
Status: Terminated | Type: Observational
Why Stopped: insufficient amount of participants
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Kenema Government Hospital (Other); London School of Hygiene and Tropical Medicine (Other); Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: 38-18
Record Dates: First submitted 2019-03-13; First posted 2019-03-26 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2019-03

CONDITIONS: Lassa Fever
MeSH Terms: conditions — Lassa Fever | interventions — Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lassa fever
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — Standard of care: Intravenous administration of ribavirin at currently recommended dosages. Loading dose of 30 mg/kg (maximum 2 g), followed by 15 mg/kg (maximum 1 g) intravenously QDS for four days, followed by 7.5 mg/kg intravenously (maximum 500 mg) TDS for six days.

SUMMARY:
Lassa fever carries a treated mortality in hospitalized patients of up to 50%. Lassa fever is often described as being characterized by vascular leak and shock in the terminal phase, but, whilst animal data supports this, there are limited data in humans. Therefore, an aim of this study therefore is to characterize cardiovascular function in patients with Lassa fever, with the ultimate goal of informing future trials of supportive or therapeutic strategies.

Ribavirin is the current standard of care. However, the efficacy of ribavirin has not been established in a randomised controlled trial (RCT). There is very limited pharmacokinetic (PK) data on ribavirin in patients with Lassa fever and the optimal dose of ribavirin for an RCT is unknown. Furthermore, there are various hypothesized mechanisms of action of ribavirin, none of which have been investigated in humans with Lassa fever. Further aims of this study therefore are to characterize the PK of ribavirin in Lassa fever, and identify any associations between ribavirin PK parameters, viral load and markers of immune/inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* Positive antigen or PCR test for Lassa fever
* Aged 10 years or above

Exclusion Criteria:

* Patients for end of life care only

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to KGH with a positive antigen or PCR test for Lassa virus.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular function - primary | Up to 28 days during hospitalisation
  Death during hospitalization
Ribavirin PK - primary | Up to 15 days during hospitalisation
  Proportion of patients with ribavirin CMIN above the IC90 at all measured CMIN during therapy
Ribavirin PD (mechanism of action) - primary | Up to 15 days during hospitalisation
  • Change in Lassa virus viral load (copies/ml) from baseline to day 3/5

SECONDARY OUTCOMES:
Cardiovascular function - secondary | Up to 28 days during hospitalisation
  • Shock (shock is defined as a systolic BP < 90mmgHg [age specific in children] OR a MAP < 65mmgHg AND a lactate > 2 mEq/L)
Cardiovascular function - secondary | Up to 28 days during hospitalisation
  • Persistent shock (persistent shock is defined as a MAP < 65 mmHg OR a SBP < 90 mmHg [age specific in children] AND a lactate > 2 mEq/L on more than 2 occasions [at least 6 hours apart] DESPITE IV fluids +/- vasopressors)
Cardiovascular function - secondary | Up to 28 days during hospitalisation
  • Respiratory distress (respiratory distress is defined as a respiratory rate > 24 (age specific in children) AND oxygen saturations < 94% OR use of supplemental oxygen)
Ribavirin PK - secondary | Up to 15 days during hospitalisation
  • Proportion of patients with ribavirin CMIN above the IC50 at all measured CMIN during therapy
Ribavirin PK - secondary | Up to 15 days during hospitalisation
  • Peak Plasma Concentration
Ribavirin PK - secondary | Up to 15 days during hospitalisation
  • Minimum Plasma Concentration
Ribavirin PK - secondary | Up to 15 days during hospitalisation
  • Area under the plasma concentration versus time curve
Ribavirin PK - secondary | Up to 15 days during hospitalisation
  • Half life
Ribavirin PD (mechanism of action) | Up to 15 days during hospitalisation
  • Change in ISG expression from baseline to day 3/5
Ribavirin PD (mechanism of action) | Up to 15 days during hospitalisation
  • Change in RHI from baseline to day 3
Ribavirin PD (mechanism of action) | Up to 15 days during hospitalisation
  • Time to negative blood PCR for Lassa virus
Ribavirin PD (mechanism of action) | Up to 15 days during hospitalisation
  • Survival to hospital discharge
Ribavirin PD (mechanism of action) | Up to 15 days during hospitalisation
  Change in aspartate aminotransferase concentrations (units/litre) from baseline to day 3/5
Ribavirin PD (mechanism of action) | Up to 15 days during hospitalisation
  • Change in systemic nitric oxide concentrations from baseline to day 3/5

CONTACTS AND LOCATIONS:
Overall Officials: Alex Salam, MD, Principal Investigator — University of Oxford
Locations (1):
- Kenema Government Hospital, Kenema, Sierra Leone

IPD SHARING:
Plan to Share IPD: Undecided